CLINICAL TRIAL: NCT03713281
Title: Evaluation of a Toric Multifocal Contact Lens Manufactured in Etafilcon Material in a Low ADD Hyperopic Population
Status: Completed | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-6278
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Visual Acuity

STUDY DESIGN:
Masking Description: Although study includes one arm, Participant is masked to the identity of the investigational product.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Test Lens (Experimental): Subjects between the ages 40 to 70 years of age and who are adapted contact lens wearers with astigmatism in both eyes will be assigned to the same Test Lens according to the lens wear schedule.
  Interventions: Device: Toric Multifocal etafilcon A with PVP

INTERVENTIONS:
Device: Toric Multifocal etafilcon A with PVP — Investigational

SUMMARY:
The study is a bilateral, single-masked, single-arm, 3-visit dispensing study. There will be one study treatment, with the subject being in the treatment for approximately 12-16 days.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be at least 40 and not more than 70 years of age at the time of screening.
  4. The subject's distance spherical component of their refraction must be in the range of +1.25 D to +3.75 D in each eye.
  5. The subject's refractive cylinder must be -1.00 to -1.50 D in each eye.
  6. The subject's ADD power must be in the range of +0.75 D to +1.50 D in each eye.
  7. Subject's refractive cylinder axis must be within 90°±30° or 180°±30° in each eye.
  8. The subject must have best corrected visual acuity of 20/20-3 or better in each eye.
  9. Subjects must own a wearable pair of spectacles if required for their distance vision.
  10. The subject must already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  7. A history of amblyopia, strabismus or binocular vision abnormality.
  8. Any current ocular infection or inflammation.
  9. Any current ocular abnormality that may interfere with contact lens wear.
  10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.
  11. Use of any ocular medication, with the exception of rewetting drops.
  12. History of herpetic keratitis.
  13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  15. Any known hypersensitivity or allergic reaction to Eye-Cept® rewetting drop solution.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Total Eye Care PA, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 30 subjects were enrolled in this study of which, 28 subjects were assigned and dispensed a study lens, while 2 subjects failed to meet all eligibility criteria. Of the total dispensed subjects, 25 completed the study and 3 subjects were discontinued.
Groups:
- Toric Multifocal Etafilcon A With PVP: All subjects that were disepnsed the sudy lens.
Period: Overall Study
Arm/Group | Toric Multifocal Etafilcon A With PVP
Started | 28
Completed | 25
Not Completed | 3
Not completed — Lens handling difficuluties | 2
Not completed — Subject was not dispensed enough lenses | 1

BASELINE CHARACTERISTICS:
Groups:
- Toric Multifocal Etafilcon A With PVP: All subjects dispensed a study lens.
Arm/Group | Toric Multifocal Etafilcon A With PVP
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.8 (4.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 3
  White | 24
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (logMAR)
Description: High Luminance, high contrast distance (4 meters) binocular visual acuity was recorded with the test contact lenses using ETDRS visual acuity charts. The logMAR visual acuity was measured as follows: 0.02 logMAR=1 letter. Where lower logMAR scores represent better vision. A value of 0.0 logMAR is equivalent to 20/20 Snellen visual acuity.
Time Frame: 2-Week Follow-up
Population: All sub jects that completed all planned study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Toric Multifocal Etafilcon A With PVP: All subjects that were dispensed the study lens.
Arm/Group | Toric Multifocal Etafilcon A With PVP
Number analyzed (Participants) | 23
logMAR | -0.13 (0.095)
Statistical Analysis 1: Comparison: Toric Multifocal Etafilcon A With PVP; Statistically superiority will be concluded if the upper confidence limit will be less than 0.10 logMAR; Test type: Superiority; Linear Mixed Model; Kenward and Roger modethod for the demoninator degrees of freedom; Least-square mean = -0.131, 95% CI 2-sided [-0.208 to -0.054], Standard Error of Mean 0.0278

2. Primary Outcome: Near Visual Acuity (logMAR)
Description: High Luminance, high contrast near (40 centimeters) binocular visual acuity was recorded with the test contact lenses using ETDRS visual acuity charts. The logMAR visual acuity was measured as follows:0.02 logMAR=1 letter. Where lower logMAR scores represent better vision. A value of 0.0 logMAR is equivalent to 20/20 Snellen visual acuity.
Time Frame: 2-Week Follow-up
Population: All subjects that completed all planned study visits without a major protocol deviation impacting a primary endpoint.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Toric Multifocal Etafilcon A With PVP
Number analyzed (Participants) | 23
logMAR | 0.06 (0.080)
Statistical Analysis 1: Comparison: Toric Multifocal Etafilcon A With PVP; Statistically superiority will be concluded if the upper confidence limit will be less than 0.17 logMAR for near distance logMAR visual acuity; Test type: Superiority; Linear Mixed Model; Kenward and Roger method for the demoninator degrees of freedom; Least-square means = 0.060, 95% CI 2-sided [-0.017 to 0.137], Standard Error of Mean 0.0278

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2 weeks per subject.
Groups:
- Toric Multifocal Etafilcon A With PVP: All subjects dispensed a stud lens.
Arm/Group | Toric Multifocal Etafilcon A With PVP
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT03713281/Prot_SAP_000.pdf